CLINICAL TRIAL: NCT00061386
Title: Reducing Disease Risk in Low Income Postpartum Women
Brief Title: Improving Health in Low Income Women Following the Birth of a Child
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01HD37368-4; 5R01HD037368 (NIH)
Record Dates: First submitted 2003-05-27; First posted 2003-05-28 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-09

CONDITIONS: Health Promotion
Keywords: Postpartum; Low income; Diet; Physical activity
MeSH Terms: conditions — Motor Activity | interventions — Nutritional Status

INTERVENTIONS:
Behavioral: Nutrition and physical activity program

SUMMARY:
This study will evaluate a community-based program to improve diet and physical activity in women during the first 12 months following the birth of a child. The program is designed to complement existing federal programs for low-income families and is directed toward low-income, postpartum, multi-ethnic women.

DETAILED DESCRIPTION:
The postpartum period is a window of opportunity to promote behaviors that reduce the risk of chronic disease and benefit reproductive health. The Expanded Food and Nutrition Education Program (EFNEP) is an educational program delivered by community-based paraprofessional's that aims to improve dietary and activity patterns among low income, multi-ethnic women during the postpartum period. This study will evaluate the efficacy of the EFNEP to impact the diet and activity patterns of women.

Women were recruited through the Special Supplemental Food Program for Women, Infants, and Children (WIC) and randomized to either the EFNEP group or a usual care group. Women in both groups will receive standard WIC care consisting of nutrition-risk and breastfeeding educational messages at postpartum and follow-up visits. Women in the EFNEP group participated in an additional two component intervention that included five home visits and motivational telephone calls from project staff.

Primary study outcomes were assessed at Months 1 and 12. Primary outcomes included fruit and vegetable intake, saturated fat intake, and physical activity. Secondary outcomes will include Body Mass Index and indicators of fat mass and distribution. The study will also analyze mediating and modifying factors, including social support and norms, perceived health status, smoking, television viewing, food insecurity, food and activity access, and utilization of federal programs and health care.

ELIGIBILITY:
Inclusion Criteria:

* Less than 20 weeks postpartum
* Receive services of USDA's Special Supplemental Food Program for Women, Infants, and Children (WIC)

Exclusion Criteria:

* Less than 18 years of age upon recruitment

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 680
Dates: Start 2001-03; Study Completion 2004-03

PRIMARY OUTCOMES:
fruit and vegetable intake
saturated fat intake
physical activity

SECONDARY OUTCOMES:
body mass index
indicators of fat mass and distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Karen E. Peterson, ScD, RD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard School of Public Health, SHDH Department, Boston, Massachusetts, United States

REFERENCES:
- [Background] Peterson KE, Sorensen G, Pearson M, Hebert JR, Gottlieb BR, McCormick MC. Design of an intervention addressing multiple levels of influence on dietary and activity patterns of low-income, postpartum women. Health Educ Res. 2002 Oct;17(5):531-40. doi: 10.1093/her/17.5.531. PMID 12408198